CLINICAL TRIAL: NCT03741920
Title: Evaluation of the Personal KinetiGraph™ (PKG™) to Improve Insight Into Parkinson's Disease Status (APPRISE)
Brief Title: Evaluation of the Personal KinetiGraph™ (PKG™) to Improve Insight Into Parkinson's Disease Status
Acronym: APPRISE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Global Kinetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Study 002
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
Keywords: Personal KinetiGraph (PKG) Movement Recording System
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Personal KinetiGraph™ (PKG™) + (Experimental): For subjects in the PKG+ Group, the study MDS will review and report on the PKG prior to the visit and use the information to guide the discussion with the subject during the clinical assessment. PKG results will be recorded in the PKG Reporting case report form (CRF). The study MDS will complete the MDS-Clinician Assessment CRF to denote patient-reported symptoms, treatable findings, and clinical management planning based on his/her routine clinical assessment procedures along with the PKG information.
  Interventions: Device: Personal KinetiGraph™ (PKG™)
- Personal KinetiGraph™ (PKG™) - (Active Comparator): For subjects in the PKG- Group (control group), the study Movement Disorder Specialist (MDS) will complete the MDS - Clinician Assessment CRF to denote patient-reported symptoms, treatable findings, and clinical management planning based on his/her routine clinical assessment procedures. The study Movement Disorder Specialist will be blinded to the PKG information until the second part of the 90-day follow-up visit.
  Interventions: Device: Personal KinetiGraph™ (PKG™)

INTERVENTIONS:
Device: Personal KinetiGraph™ (PKG™) — The Personal KinetiGraph™ (PKG™) Movement Recording System was developed by neurologists at the Melbourne-based Florey Institute of Neuroscience and Mental Health. The product is manufactured and marketed by Global Kinetics (GKC).
  The Personal KinetiGraph™ (PKG™) Movement Recording System consists of the following:
  * A wrist-worn data logger designed to acquire data on the kinematics of movement disorder symptoms over a 6-10 day period.
  * An application to configure the data logger and transfer the acquired data at the end of a recording.
  * A series of algorithms that analyze the uploaded data, producing a report that is delivered to the clinician. The report contains objective data distinguishing the movement patterns consistent with tremor, bradykinesia, dyskinesia and immobility.

SUMMARY:
The primary objective is to understand the utility of Personal KinetiGraph movement recording system data in the clinical management of Parkinson's disease (PD) in routine clinical care at a movement disorders clinic. Specifically:

1. Measure medication use and clinical management plan changes in a large, multicenter cohort among participants undergoing a clinical assessment with an MDS in which the MDS reviews the participant's PKG during the clinical assessment in half of the enrolled participants (PKG + Group) and in half of the enrolled participants the MDS completes the clinical assessment without the PKG (PKG- Group).
2. Determine the association between frequency of medication changes, the PKG information, and other clinical assessments among participants with and without a PKG report of their PD motor status available to the clinician at the time of evaluation.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled trial. The study consists of 3 phases as follows:

* Randomization phase: subjects undergo screening, baseline, interim and 90-day follow-up visits

  * PKG+ Group (standard of care clinical evaluation plus use of PKG data)
  * PKG- Group (standard of care clinical evaluation without use of PKG data - the MDS is blinded to PKG data)
  * Randomization ratio will be 1:1 with assignments generated in advance of the start of the trial by the unblinded statistician who will provide a list containing group assignments that will be available in an Electronic Database (EDC) for site use.
  * The clinical investigator, study site staff, and subject will not be blinded to the randomization assignment during the randomization phase of the study
* Open-label phase: at the end of the 90-day randomization phase visit for PKG- Group subjects, the MDS will report on the PKG and review it with the subject, the subject will complete follow-ups with the MDS using the PKG information during the clinical assessment following the same process as the PKG+ Group during the randomization phase
* Extended open-label follow-up phase: annual follow-ups for all subjects at 1, 2, and 3 years during which the MDS will use the PKG information during clinical assessments for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign a written informed consent for study participation
* Age 46 - 83 years at the time of consent (per PKG Indications for Use, see Technical Instructions Manual)
* Responsive to dopaminergic medications

Exclusion Criteria:

* Contraindication to increasing dopaminergic therapy, such as current or treated freezing gait, symptomatic postural hypotension, or bothersome hallucinations
* Wheelchair bound or bedridden
* Utilizing or planning advanced PD therapies (DBS, infusion, etc.)
* History of delirium in the past year
* In the investigator's or sponsor's opinion, subject has any unstable or clinically significant condition that would impair the participant's ability to comply with study requirements or interfere with interpretation of the study endpoints (e.g., subject able to complete PKG wear instructions per Patient Instruction Manual, or ability to comply with required study procedures and visit schedule)

Ages: 46 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment changes with or without the use of PKG data | 90 day
  The proportion of patients in which the clinical management plan was changed in patients followed in the PKG- Group (clinician standard of care) compared to the PKG+ Group (clinician standard of care with the use of PKG data).

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Pahwa, MD, Principal Investigator — University of Kansas Medical Center
Locations (12):
- United States (12):
  - Sutter Health, Sacramento, California
  - University of California, San Diego, California
  - Parkinson's Disease and Movement Disorders Center, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Medical Institute, Baltimore, Maryland
  - Michigan State University, East Lansing, Michigan
  - Northwell Health, Great Neck, New York
  - New York University, New York, New York
  - University of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maetzler W, Klucken J, Horne M. A clinical view on the development of technology-based tools in managing Parkinson's disease. Mov Disord. 2016 Sep;31(9):1263-71. doi: 10.1002/mds.26673. Epub 2016 Jun 7. PMID 27273651
- [Background] Pahwa R, Isaacson SH, Torres-Russotto D, Nahab FB, Lynch PM, Kotschet KE. Role of the Personal KinetiGraph in the routine clinical assessment of Parkinson's disease: recommendations from an expert panel. Expert Rev Neurother. 2018 Aug;18(8):669-680. doi: 10.1080/14737175.2018.1503948. Epub 2018 Jul 26. PMID 30032695
- See also: Related Info — https://www.globalkineticscorporation.com/